CLINICAL TRIAL: NCT05068128
Title: Combined Flow-pressure Study of Cerebrospinal Circulation Using CSF Perfusion Tests and Phase-contrast MRI - Reversible Dementia Substudy
Brief Title: Combined Flow and Pressure Study of Craniospinal Dynamic
Acronym: REVERT
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: University Hospital, Caen (Other); University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0017
Record Dates: First submitted 2021-09-07; First posted 2021-10-05 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Intracranial Pressure; Cerebral Blood Flows; Infusion Test; Phase Contrast MRI; Hydrocephalus; Dementia
Keywords: Intracranial pressure; cerebral blood flows; infusion test; Phase contrast MRI; Hydrocephalus; Dementia
MeSH Terms: conditions — Hydrocephalus; Dementia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Flow MRI — 4 flow acquisitions based on the 2D cine phase contrast sequence (present on all MRI systems) will be performed.
  This sequence requires a cardiac synchronization by a plethysmograph put on the patient's finger.
  32 cardiac phases are reconstructed per acquisition. The processing of the flow MRIs and the analysis of the flow curves of the LCS and blood during the cardiac cycle will be performed using the Amiens software.
  Parameters measured via flow MRI are:
  - Cerebral vascular flow, intracranial LCS dynamic volume, extracranial LCS dynamic volume
Other: PERFUSION TEST — The test will be performed will include:
  * Inserting a needle into the lumbar space, Ommaya reservoir or valve pre-chamber, as appropriate
  * Connect the needle to the pressure transducer via saline filled manometer lines connected via a 3-way valve. The other end of the 3-way connection will be connected to a saline
  * Recording of the opening pressure for 10 minutes
  * The infusion test is terminated either when the pressure stabilizes again on a new plateau, or when the average pressure exceeds 40 mmHg, or in case of adverse effects or symptoms such as headache, nausea/vomiting or visual disturbances.
  * At the end of the test, a depletion of 30 to 50 mL of CSF will be performed.
  * The pressure recording during the test is then used to calculate the parameters of the mechanical properties of the CSF circulation and reported to the neurosurgeon ordering the test.

SUMMARY:
Normal pressure hydrocephalus (NPH) can cause a type of dementia. However, this type of dementia is the only one that is reversible. To treat this dementia it is necessary to evacuate the accumulation of CSF from the brain to another body cavity using a device called a shunt. But the implantation of this shunt is only effective when the cause of the pathology is an alteration of the normal circulation of the CSF. To diagnose these patients, morphological MRI and lumbar puncture are standard approaches used but remain perfectible in diagnostic terms.

The main objective is to build a new model of the interaction of intracranial pressures and fluids in order to obtain a new parameter allowing to obtain information on the cerebral biomechanics.

ELIGIBILITY:
Inclusion Criteria:

* age > 55 years
* Patients with suspected active hydrocephalus (HA) known as "normal pressure":
* Ventricular dilatation: Evans index > 0.3
* Patients with cognitive impairment, and/or gait disorders and/or urinary incontinence or a combination of these three symptoms.
* Absence of other neurological diseases that could cause ventriculomegaly.
* Information and collection of the patient's non opposition

Exclusion Criteria:

* All patients with neurological disease other than active hydrocephalus will be excluded.
* Individuals who cannot tolerate an MRI examination
* All individuals with implants, pacemakers, prostheses and ferromagnetic objects
* Patients under guardianship, curators or safeguard of justice

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected active hydrocephalus (HA) known as "normal pressure" and with Flow MRI and CSF infusion test.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Variation of number of MRICP parameters according of CSF accumulation | up to 3 years
  The MRICP parameter will combine the CSF pressure and CSF flows. MRICP parameter results of the interaction of intracranial pressures and fluids in order allowing to obtain information on the cerebral biomechanics.
  Accumulation of CSF from the brain to another body cavity is neccessary to be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Salouël, France

IPD SHARING:
Plan to Share IPD: No